CLINICAL TRIAL: NCT00080574
Title: The Effects of Thyroid Hormone on Cytochrome P450 and P-Glycoprotein Activity in Thyroid Cancer Patients
Brief Title: The Effect of Thyroid Hormone on Drug Elimination in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040140; 04-DK-0140
Record Dates: First submitted 2004-04-07; First posted 2004-04-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Thyroid Cancer
Keywords: Pharmacokinetics; Drug Metabolism; Levothyroxine; Hypothyroidism; Hyperthyroidism; Drug Interactions; Cytochrome P450; P-Glycoprotein; Drug Transport Proteins; Thyroid Hormone; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Hypothyroidism; Hyperthyroidism

INTERVENTIONS:
Procedure: Skin Biopsy

SUMMARY:
This study will examine whether and how levothyroxine (Synthroid, a synthetic thyroid hormone) affects the way the body handles other drugs. If levothyroxine does affect the metabolism of other drugs, the dose of those medications may need to be increased to enhance their action or decreased to avoid adverse reactions.

Patients 18 years of age and older with thyroid cancer who are participating in NIH protocol #77-DK-0096 and are receiving long-term suppression therapy with levothyroxine may be eligible for this study. This is not a study of thyroid cancer or of potential new drugs to treat it. Thyroid cancer patients are being studied because their treatment regimen provides an opportunity to study drug metabolism while patients are both on and off levothyroxine therapy.

Participants come to the NIH Clinical Center on two occasions: once while they are regularly taking their levothyroxine, and once while they are off the medication in preparation for their radioactive iodide diagnostic scan for the procedures outlined below. The time interval between the two clinic visits depends on whether the first visit is while the patient is on or off medication. Participants are asked to fast overnight before each visit and to abstain from certain foods and beverages for 48 to 72 hours before the visit. At each visit, patients undergo the following procedures:

* Medication history, limited physical examination, and blood draw for laboratory tests, including a test to look for genes important in eliminating medications from the body.
* Insertion of a catheter (thin plastic tube) into an arm vein for collecting blood samples.
* Shave skin biopsy (optional) to explore how proteins in the skin that metabolize and transport drugs are affected by thyroid hormone. For this procedure, the skin is cleaned, numbed with medicine, and a small sample of the top layer is removed with a razor blade. The wound heals in 2 to 3 days.
* Medication dosing. Participants take all of the following substances by mouth at the same time: 1) 200 mg of caffeine, a compound commonly found in chocolate, soda/pop, coffee, tea and non-prescription products to prevent sleep; 2) 30 mg of dextromethorphan, a non-prescription cough suppressant; 3) 40 mg of omeprazole, a prescription drug for heartburn and stomach ulcers; 4) 8 mg of midazolam, a prescription drug used to cause relaxation and drowsiness; and 5) 120 mg of fexofenadine, a non-sedating prescription antihistamine used to treat allergies.
* Blood and urine sampling. Fifteen blood samples of about 5 mL (1 teaspoon) each are collected through the catheter and urine is collected over the next 24 hours to determine what happens to the test drugs in the body.

Participants may resume their normal diet 4 hours after taking the study medications.

DETAILED DESCRIPTION:
Interaction between thyroid hormones and commonly prescribed drugs has been well documented, resulting in augmentation or attenuation of the action of either compound. Phase I drug metabolism is mediated mostly by enzymes belonging to the cytochrome p450 superfamily. Studies in animals and cell cultures have shown that thyroid hormones play an important role in the constitutive expression of the p450 enzymes, thus potentially altering the metabolism and the effects of a variety of drugs. P-glycoprotein is expressed in the major organs associated with drug absorption, distribution, and elimination from the body (e.g. intestine, kidney, liver, skin, and the blood-brain barrier). Expression of intestinal P-glycoprotein in humans also appears to be influenced by thyroid hormones. We intend to study the effect of thyroid hormones on the activity of CYP1A2, CYP2C19, CYP2D6, CYP3A4 and P-glycoprotein by using a five-drug cocktail (caffeine, omeprazole, dextromethorphan, midazolam, and fexofenadine) administered in patients with thyroid cancer, both on thyroid hormone suppression therapy (in conditions of subclinical hyperthyroidism) and off this treatment (in conditions of hypothyroidism) at the time of their routine radioactive iodine scan. Additionally we will perform two skin biopsies in order to assess the pattern of expression of metabolic enzymes and drug transport proteins on and off thyroid hormone suppression therapy.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subject has signed the informed consent document;
2. Subject is greater than or equal to 18 years of age;
3. Subjects diagnosed with thyroid cancer participating in protocol 77DK0096;
4. Subjects receiving THST with levothyroxine;
5. Serum TSH less than 0.4 mIU/L while on THST, and more than 20 mIU/L while off THST.

EXCLUSION CRITERIA:

Subject is pregnant, currently breast-feeding, practicing birth control with hormonal contraceptives, or is on hormone replacement therapy (HRT).

Subject is a smoker.

Subject has a confounding medical illness (es) that in the judgement of the investigators would pose an added risk for the subject (e.g. severe respiratory disease).

Subject has a history of substance abuse within the past 5 years or drug or alcohol use, that may affect enzyme levels and function.

Caffeine or caffeine-containing beverages and chocolate bars consumption within 48 hours of scheduled caffeine administration for CYP1A2 phenotyping; scheduled omeprazole administration during or within 14 days of the study; scheduled dextromethorphan administration during or within 30 days of study; scheduled fexofenadine administration during or within 7 days of the study.

AST or ALT greater than or equal to 2 times the upper normal reference limit.

Concurrent administration of known CYP and/or P-gp inducers (barbiturates, phenytoin, carbamazepine, rifampicin) and inhibitors (amiodarone, atorvastatin, chloroquine, cimetidine, co-trimoxazole, cyclosporine, diltazem, erythromycin, fluoxetine fluvoxamine, isoniazid, itrakonazole, ketokonazole, metronidazole, mexiletine, nefazadone, norfloxacin, verapamil) or use of any alternative/complementary therapies for at least 30 days prior to study or during the study. Non-herbal vitamin and mineral preparations will be allowed.

Inability to obtain venous access for sample collection, or basal hemoglobin of equal or less than 10 g/dl.

Patients receiving scheduled therapy with alprazolam, triazolam, clonazepam, diazepam, lorazepam, oxazepam, temazepam or chlorodiazepoxide, during or within 30 days of study.

Patients consuming grapefruit products (juice or the fresh fruit), apple and orange juice during or within 72 hrs of study.

History of intolerance to caffiene, omeprazole, dextromethorphan, midazolam or fexofenadine.

The presence of persistent diarrhea or malabsorption syndromes that would interfere with the patient's ability to adequately absorb drugs; and/or

Patients receiving monoamine oxidase inhibitors (MAOIs) such as phenelzine, tranylcypromine, and isocarboxazid.

Patients with a history of cheloids formation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-04; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Meisel C, Gerloff T, Kirchheiner J, Mrozikiewicz PM, Niewinski P, Brockmoller J, Roots I. Implications of pharmacogenetics for individualizing drug treatment and for study design. J Mol Med (Berl). 2003 Mar;81(3):154-67. doi: 10.1007/s00109-002-0417-4. Epub 2003 Mar 15. PMID 12682724
- [Background] Nolan SR, Self TH, Norwood JM. Interaction between rifampin and levothyroxine. South Med J. 1999 May;92(5):529-31. doi: 10.1097/00007611-199905000-00018. PMID 10342905
- [Background] Blackshear JL, Schultz AL, Napier JS, Stuart DD. Thyroxine replacement requirements in hypothyroid patients receiving phenytoin. Ann Intern Med. 1983 Sep;99(3):341-2. doi: 10.7326/0003-4819-99-3-341. No abstract available. PMID 6614682